CLINICAL TRIAL: NCT05659043
Title: The Impact of Glycation Modification of apoA-I on HDL Function and Atherogenesis in Type Diabetes Mellitus
Brief Title: Glycation of apoA-I and Diabetic Atherogenesis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 81870357
Record Dates: First submitted 2022-12-11; First posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma and PBMCs
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- T2DM with CAD: Diagnosis of T2DM was made according to the criteria of the American Diabetes Association. The patients were tested by angiography, with CAD diagnosed if luminal diameter narrowing was estimated visually at ≥50% in a major epicardial coronary artery.
  Interventions: Other: overnight fasting
- T2DM without CAD: Diagnosis of T2DM was made according to the criteria of the American Diabetes Association. These subjects had no history of ischemic heart disease (acute myocardial infarction, unstable angina, chronic stable angina, previous percutaneous or surgical coronary revascularization, heart failure) and received CCTA in the outpatient clinics due to suspected CAD or other causes. And the luminal diameter narrowing was estimated by CCTA at ≤30%.
  Interventions: Other: overnight fasting

INTERVENTIONS:
Other: overnight fasting — All blood samples were taken on the day of cardiac catheterization after overnight fasting.

SUMMARY:
The goal of this study is to determine the relationship of apoprotein A-1 (apoA-I) glycation and development of diabetic atherosclerosis.

ApoA-I is crucial for reverse cholesterol transport and anti-inflammation/anti-atherosclersis functions of HDL. However, apoA-I is easily subjected to non-enzymatic glycation modification in diabetic milleu. Our preliminary study has shown that apoA-I in HDL from type 2 diabetes mellitus (T2DM) patients with coronary artery disease (CAD) is significantly glycated, and site specific glycation of apoA-I impairs HDL function and is related to the development of atherosclerosis. To the best of our knowledge, less clinical information regarding apoA-I glycation and CAD has been reported. In this cross-sectional study, by consecutively enrolling diabetic patients with (two to three hundred) or without CAD (controls, six to eight hundred) in our hospital, we will isolate their serum HDL and perform a qualitative and quantitative proteomic analysis of apoA-I glycation. The relation of apoA-I glycation and HDL function and angiography-determined severity of CAD will be evaluated. Later, we will follow these diabetic patients to analyze the influence of apoA-I glycation on the outcome including plaque progression.

DETAILED DESCRIPTION:
The goal of this study is to determine the relationship of apoprotein A-1 (apoA-I) glycation and development of diabetic atherosclerosis.

ApoA-I is crucial for reverse cholesterol transport and anti-inflammation/anti-atherosclersis functions of HDL. However, apoA-I is easily subjected to non-enzymatic glycation modification in diabetic milleu. Our preliminary study has shown that apoA-I in HDL from type 2 diabetes mellitus (T2DM) patients with coronary artery disease (CAD) is significantly glycated, and site specific glycation of apoA-I impairs HDL function and is related to the severity of atherosclerosis. To the best of our knowledge, less clinical information regarding apoA-I glycation and CAD has been reported. In this cross-sectional study, we will consecutively enroll several hundred diabetic patients (two to three hundred) with no CAD (less than stenosis of 25% in coronary CTA) as controls. And we will also consecutively enroll several hundred (six to eight hundred) angiographically established T2DM patients with CAD (stenosis of >50% in coronary angiography). Serum HDL of all participants will be isolated and a qualitative and quantitative proteomic analysis of apoA-I glycation will be performed by mass spectrometry. The relation of apoA-I glycaiton and HDL function and angioraphy-determined severity of CAD will be evaluated. Later, we will follow these diabetic patients for approximately two years to analyze the influence of apoA-I glycation on the clinical outcomes (stroke, myocardial infarction, hospitalization for heart failure, death due to cardiovascular causes, etc) including plaque progression.

ELIGIBILITY:
Inclusion Criteria:

Type 2 diabetes diagnosed by one of the following criteria:

HbA1c >/= 6.5% Fasting plasma glucose >/= 7.0 mmol/l (confirmed) 2h plasma glucose value during OGTT >/= 11.1 mmol/l Already receiving glucose-lowering agents; Receiving coronary angiography for clinically suspected CAD (T2DM with CAD), Receiving CCTA for suspected CAD or other causes (T2DM without CAD).

Exclusion Criteria:

Severe liver failure (Child-Pugh grade B to C)； Severe anemia (hemoglobin < 60g/L)； Familial hypercholesterolemia； Active malignant tumor； Active autoimmune diseases on corticosteroids； Acute or chronic infection； Death.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is a single-center cohort study. Patients with type 2 diabetes and suspected coronary artery disease undergone coronary angiography at Ruijin Hospital, Shanghai, China are consecutively enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Qualitative and Quantitative Mapping ApoA-I Glycation Modification Profiles | completion date - December 2021
  One of aims is understanding the importance of apoA-I glycation modification in HDL dysfunction and the progression of diabetic CAD, a comprehensive analysis of apoA-I glycation modification requires numerous levels of information, including (1) the type of glycation modification, (2) glycation localization, (3) glycation frequency in the subject cohort, and (4) the extent of glycation. The other aim is identifying the crucial pathogenic glycation sites of apoA-I based on apoA-I glycation modification profiles. Defining the chemistry of the pathologic glycation sites of apoA-I during progression of CAD will allow us to target specific epitopes using therapeutic antibodies or small molecules at every stage of disease.

SECONDARY OUTCOMES:
Individual ApoA-I Glycation Profiles Variability and Cardiovascular Events | December 2023
  Individual ApoA-I Glycation Profiles Variability is evaluated annually，and The incidence of MACCE (major adverse cardio and cerebral vascular events), lesion associated events (target lesion myocardial infarction, target lesion faliure, target vessel Revascularization, etc. observed continuously for 3 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided